CLINICAL TRIAL: NCT07158853
Title: Combined tDCS and Cognitive Training as an Adjunctive Treatment in Opioid Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYCH-2025-34164
Record Dates: First submitted 2025-08-11; First posted 2025-09-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Opioid Use Disorder; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Soterix Mini-CT Remote tDCS systems offer fully reliable researcher and participant blinding. Soterix Mini-CT Remote tDCS software interface allows for automatic generation of sham versions of the protocol. The system is run with a password-protected mode - minimizing information presented on the screen for definitive blinding of research staff and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- tDCS (Active Comparator): All intervention sessions will use the Soterix Mini-CT Remote tDCS device
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham Electrodes (Placebo Comparator)
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — We will deliver 2-mA tDCS current intensity during a 30 minute stimulation period (including a 30-second ramp-up and 30-second ramp-down period) to the dorsolateral prefrontal cortex. Electrodes will be fixed on marked locations based on the 10-20 EEG system. Anodal stimulating electrode will be over the left DLPFC (F3) and cathodal electrode over the right DLPFC (F4).
  Arms: tDCS
Device: Sham Stimulation — electrodes will have the same montage as active tDCS (F3/F4), but current will be ramped down after the initial 30 seconds ramp-up period. Thus, participants will feel the initial sensation associated with tDCS but will receive no active current for the rest of the stimulation period.
  Arms: Sham Electrodes

SUMMARY:
The overall goal of this study is to investigate the added benefit of a neuromodulation intervention in individuals under buprenorphine maintenance treatment for OUD (bOUD).

ELIGIBILITY:
Inclusion Criteria:

* ability to provide consent and comply with study procedures
* Diagnostic and Statistical Manual of Mental Disorders criteria for OUD
* undergoing buprenorphine maintenance treatment. Participants may have current comorbid drug use, but primary diagnosis must be OUD
* Intention to remain in the addiction treatment program until intervention completion.

Exclusion Criteria:

* Any medical condition with neurological sequelae
* head injury resulting in skull fracture or loss of consciousness of >30 minutes
* any tDCS or MRI contraindication (tDCS: history of seizures, metallic cranial plates/screws or implanted device, history of eczema on scalp. MRI: unapproved metallic implants, pacemakers or any other implanted electrical device, shrapnel, metallic braces, non-removable body piercings, pregnancy, breathing or movement disorder, or claustrophobia)
* any psychotic disorder (participants with other treated and stable psychiatric disorders will be included)
* presence of a condition that would render study measures impossible to administer or interpret
* age younger than 18
* primary current substance use disorder on a substance other than opioids except for caffeine or nicotine
* court mandated treatment
* pregnancy
* disrespectful behavior towards the investigators and staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-04 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
tDCS effect on circuit-based target engagement of a prefrontal-incentive salience network | immediately after the intervention
  Compare change in correlation value (which represents the functional connectivity between pre-frontal cortex and prefrontal-incentive salience network) via paired t-test, from pre- to post-intervention
tDCS effect on executive functioning | immediately after the intervention
  Compare change in mean cognitive performance via paired t-test from pre-intervention cognitive assessment to post-intervention cognitive assessment (post-intervention mean cognitive score minus pre-intervention mean cognitive score) between active tDCS and sham groups

CONTACTS AND LOCATIONS:
Overall Officials: Jazmin Camchong, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No